CLINICAL TRIAL: NCT05506254
Title: A Long-term Follow-up Study of Patients in LogicBio Clinical Trials for Methylmalonic Acidemia Characterized by MMUT Mutations Who Received hLB-001
Brief Title: Long-term Follow-up Study of Patients Who Received hLB-001 Gene Therapy
Status: Active, not recruiting | Type: Observational
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: LB-001LT
Record Dates: First submitted 2022-08-16; First posted 2022-08-18 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Methylmalonic Acidemia
MeSH Terms: conditions — Methylmalonic acidemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who have previously received hLB-001
  Interventions: Drug: hLB-001

INTERVENTIONS:
Drug: hLB-001 — hLB-001 gene therapy

SUMMARY:
This is a non-interventional long-term follow-up study of patients who have participated in LogicBio studies for the treatment of MMA and received hLB-001

DETAILED DESCRIPTION:
Patients will be followed for a period of 15 years which includes the duration of time that the patient was in the treatment study.

ELIGIBILITY:
Inclusion Criteria:

* Participant has previously participated in a LogicBio clinical trial and received hLB-001.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a non-interventional long-term follow-up study of participants who have participated in LogicBio studies for the treatment of MMA and received hLB-001.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2022-07-15 (Actual); Primary Completion 2037-01-01 (Estimated); Study Completion 2037-01-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events | 15 years

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Clinical Trial Site, Atlanta, Georgia
  - Clinical Trial Site, Pittsburgh, Pennsylvania
  - Clinical Trial Site, Nashville, Tennessee
  - Clinical Trial Site, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided